CLINICAL TRIAL: NCT06532045
Title: Effect of Transcutaneous Electrical Nerve Stimulation on Patients With Palmar Hyperhidrosis
Brief Title: Effect of TENS on Patients With Palmar Hyperhidrosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Boring and feared
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed, Professor doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004611
Record Dates: First submitted 2024-07-18; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Hyperhidrosis Primary Focal Palms
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TENS arm (Experimental): This arm who was experimental group who received transcutaneous electrical nerve stimulation and breathing exercises
  Interventions: Device: Transcutaneous electrical nerve stimulation
- Breathing arm (Sham Comparator): This arm was sham and not received official treatment
  Interventions: Device: Transcutaneous electrical nerve stimulation

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation — TENS applied for 30 min for each time, five times a week, for 2 weeks and deep breathing relaxation exercise given to the intervention group twice a day (10min/exercise) for two weeks.
  Other Names: TENS

SUMMARY:
To investigate the effectiveness of Transcutaneous Electrical Nerve Stimulation on Hyperhidrosis Severity on patients with primary Palmar Hyperhidrosis.

DETAILED DESCRIPTION:
Hyperhidrosis might be a primary condition or secondary condition due to medications or systemic disorders. Primary hyperhidrosis is usually focal,bilateral, and symmetric. It mainly affects the axillae, palms, soles, face, and scalp. The incidence of primary hyperhidrosis has been reported to be between 0.6%~2.8% in both genders. Symptoms usually begin in childhood or around puberty. It interferes with daily social and occupational activities of patients and significantly impacts their quality of life.

Various treatments have been proposed to control primary hyperhidrosis. The treatment options for hyperhidrosis include topical therapy, anticholinergic, iontophoresis, botulinum toxin and surgery.

In addition to these treatment options for hyperhidrosis, several medical devices delivering energy to destroy sweat glands are undergoing promising clinical investigation. Microwave technology, several lasers (such as 1,064-nm, 1,320-nm, and 1,440-nm neodymium: yttrium- aluminum-garnet laser, 924-nm and 975-nm diode laser, long-pulsed 800- nm diode laser), micro needle radio frequency, and ultrasound technology could be included as example of the device.

In spite of these treatment options, the best therapeutic choice is still undefined. This concept encourages us to investigate the effectiveness of recent technique in the current research.

Up till now, the available literatures show a gap in knowledge and lack of well-designed studies. We will concern on the effect of Transcutaneous Electrical Nerve Stimulation on Hyperhidrosis Severity on patients with primary Palmar Hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* • Age range from 18 to 30 years old.

  * Patients will be from both sexes.
  * Body mass index from 18.5 to 24.9
  * Subject suffer from primary palmar hyperhidrosis.
  * No clinical treatment for palmar hyperhidrosis within the past month.

Exclusion Criteria:

* • Patients outside the target range.

  * Patients who were pregnant or lactating.
  * Patients who had metal implants such as a pacemaker.
  * Patients who had history of ischemic heart disease or arrhythmias.
  * Patients who had any other diseases that could be the cause ofsecondary hyperhidrosis.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Change the severity of hyperhidrosis | 2 weeks
  Measure the rate sweating by iodine starch testin unit of score

SECONDARY OUTCOMES:
Change the quality of life | 2 weeks
  Measure Quality of life by questionnaire in unit of grade

CONTACTS AND LOCATIONS:
Overall Officials: Amir Saleh, Professor, Principal Investigator — Cairo University
Locations (1):
- Mahmoud, Cairo, Cairo Government, Egypt